CLINICAL TRIAL: NCT00669006
Title: National Neuropathic Pain Database Study
Brief Title: Neuropathic Pain Database
Acronym: NePDatabase
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canada Foundation for Innovation (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: R-07-835; 13930E
Record Dates: First submitted 2008-04-28; First posted 2008-04-29 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-02

CONDITIONS: Neuropathic Pain
Keywords: neuropathic pain; database; prospective; national
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: New patients with a diagnosis of Neuropathic Pain

SUMMARY:
To establish the infrastructure for a national neuropathic pain database.

To determine the longterm outcome of the management of chronic neuropathic pain including pain relief, disability, and quality of life.

DETAILED DESCRIPTION:
The database will provide standard information on demographics, diagnosis, treatment interventions and outcome modeled on guidelines from the expert panel on initiatives on Methods, Measurement and Pain Assessment in Clinical Trials (IMMPACT)(Turk et al.,Pain 2003;106:337-345) The IMMPACT panel determined that patients should be evaluated according to six core domains as follows: Pain, physical functioning, emotional functioning, subject rating of global satisfaction with treatment, symptoms and adverse events and subject disposition.

The database will allow us to examine outcomes based on single (eg. pregabalin) and multiple (e.g tricyclic antidepressants and gabalin) therapeutic interventions. Standard guidelines for management of neuropathic pain acknowledge that polypharmacy is appropriate when individual first line treatments fail to provide adequate pain relief (Gilron I et al., CMAJ 2006; 175: 265-275; Attal N et al., European Journal of Neurology 2006; 13: 1153-1169)

ELIGIBILITY:
Inclusion Criteria:

* Primarily Neuropathic Pain
* Able to give informed consent
* Estimated Life Expectancy of 2 years

Exclusion Criteria:

* Not primarily neuropathic pain
* Declined participation- too much traveling
* Declined participation- Unknown
* Declined participation- Other, specify
* Considered unreliable- personality disorder
* Considered unreliable- cognitive impairment
* Considered unreliable- substance abuse
* Considered unreliable- Other
* Language barrier
* Exceeded quarterly quota
* Presentation with progressive or recurrent cancer, fibromyalgia, perineal pain of unknown etiology
* Other, specify

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New patients referred to the outpatient pain clinic with a diagnosis of Neuropathic Pain.
Sampling Method: Probability Sample
Enrollment: 789 (Actual)
Dates: Start 2008-04; Primary Completion 2012-02 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
To establish the infrastructure for a national Neuropathic Pain Database. | 2 years
  To establish the infrastructure for a National Neuropathic Pain Database, with a composite primary outcome measure in average pain intensity (based on average pain intensity of BPI) and reduction in disability (based on Interference Scale Score of BPI))

SECONDARY OUTCOMES:
To determine the longterm outcome of the management of chronic neuropathic pain including pain relief, disability and quality of life. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Moulin, MD, Principal Investigator — London Health Sciences Centre- St. Joseph's Health Care
Locations (1):
- London Health Sciences Centre- St. Joseph's Health Care, London, Ontario, Canada